CLINICAL TRIAL: NCT04079881
Title: Glucagon Response to Prandial Insulin Administration in Persons With Type 1 Diabetes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 201909013
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Type 1 Diabetes; Hyperglycemia, Postprandial
Keywords: glucagon; post-prandial glucose; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned receive intervention A then intervention B or to receive intervention B than intervention A
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Pre-prandial insulin administration) : B (post-prandial insulin administration) (Experimental): VISIT 1: Pre-prandial insulin: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal.
  Then VISIT 2: Post-prandial insulin: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min post the meal.
  Interventions: Drug: Insulin
- B (post-prandial insulin administration) : A (Pre-prandial insulin administration) :b (Experimental): VISIT 1: Post-prandial insulin: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min post the meal.
  Then VISIT 2: Pre-prandial insulin: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
  Other Names: Pre-prandial insulin; postprandial insulin

SUMMARY:
Glucagon regulation and response in persons with T1D at the basal state and in response to various stimuli remains unclear. Dr. Philip Cryer has previously reported that, in T1D young adults with a course of the disease of 16+9 years, the absence of endogenous insulin secretion results in increased glucagon secretion after a mixed meal, concluding that endogenous insulin reciprocally regulates the alpha-cell glucagon secretion and also suggesting that glucagon dysregulation may play an important role in post-prandial hyperglycemia in T1D. Interestingly, recent research on human islets have shown that insulin inhibits counter-regulatory glucagon secretion by a paracrine effect mediated by SGLT2-dependent stimulation of somatostatin release. An important gap in our knowledge is whether the timing of prandial insulin doses affects the glucagon response to a hyperglycemic stimulus in patients with T1D who have undetectable C-peptide.

Whether appropriately timed exogenous insulin can modify the glucagon response to glucose fluctuations has not been studied. As such, this pilot study aims to characterize the glucagon response to meal-time hyperglycemia and to compare the difference in glucagon secretion when mealtime bolus insulin is given before the meal versus after the meal with the objective of understanding factors that contribute to the peak post-prandial blood glucose and AUC of blood glucose after a mixed meal in this target population.

DETAILED DESCRIPTION:
Glucagon regulation and response in persons with T1D at the basal state and in response to various stimuli remains unclear. Dr. Philip Cryer has previously reported that, in T1D young adults with a course of the disease of 16+9 years, the absence of endogenous insulin secretion results in increased glucagon secretion after a mixed meal , concluding that endogenous insulin reciprocally regulates the alpha-cell glucagon secretion and also suggesting that glucagon dysregulation may play an important role in post-prandial hyperglycemia in T1D. Interestingly, recent research on human islets have shown that insulin inhibits counter-regulatory glucagon secretion by a paracrine effect mediated by SGLT2-dependent stimulation of somatostatin release. An important gap in our knowledge is whether the timing of prandial insulin doses affects the glucagon response to a hyperglycemic stimulus in patients with T1D who have undetectable C-peptide.

T1D course. In general, loss of 80% of beta cell function is needed to develop severe hyperglycemia. Endogenous insulin secretion is almost entirely lost within 3 to 5 years after the diagnosis . In children with new diagnosis of T1D, glucagon levels were highly associated with post prandial blood glucose, but not with HbA1c level. It has also been reported that postprandial hyperglucagonemia worsens significantly while C-peptide secretion declines during the first year of the disease. Also, in children with greater than five years of T1D, postprandial glucagon levels increased 160% from one to sixty months after diagnosis (8) and in those with disease duration of 6.9 + 4 years, glucagon levels were strongly correlated with post-prandial glucose and mildly correlated with HbA1C levels. A study in T1D adults performed in China showed that post-prandial glucagon levels were higher in T1D patients in the first year of the disease compared to those with longer course of the disease, and that hypoglycemic events were lower in newly diagnosed patients, suggesting that glucagon secretory function may become impaired with longer duration of the disease. These studies suggest that glucagon dysregulation could impact glucose control with exogenous insulin, and that this dysregulation may change with disease duration.

Post-prandial hyperglycemia adds to glucose variability, difficulty with insulin dosing and overall instability of glucose control. A recent analysis from the T1D Exchange study, that included 4768 participants younger than 26 years with a clinical diagnosis of T1D for at least 1 year showed that 21% of the participants reported administering insulin several minutes before, 44% immediately before, 10% during, and 24% after meal. Interestingly, participants who reported administering insulin during or after a meal were more likely to report missing ≥1 mealtime insulin dose per week compared with those who administered insulin before meals. In addition, a sub-analysis showed that participants who dose mealtime insulin in the postprandial period have poorer glycemic control and greater frequency of severe hypoglycemia. However, despite of these recent results, patients are often advised to give insulin after eating because caloric intake is uncertain. Understanding the mechanisms behind the higher post-prandial peak in glucose with delayed insulin administration may help clinicians guide appropriate timing of insulin administration for T1D patients with long course of the disease.

Glucagon Regulation:

Different models have been used to study glucagon regulation. Since both hyperglycemia and hypoglycemia stimulate alpha cells to produce glucagon, both the lack of intra-islet insulin and this U-shaped glucagon response contribute to glucose dysregulation in T1D . It has been reported that in T1D patients with a duration of the disease of 26.4+7.5 years, glucagon levels increased in response to the OGTT under euglycemic and hyperglycemic conditions, however the relative contribution of hyperglucagonemia to post-prandial glucose rise in the presence or absence of preprandial insulin has not been clearly elucidated. Whether appropriately timed exogenous insulin can modify the glucagon response to glucose fluctuations has not been studied. As such, this pilot study aims to characterize the glucagon response to meal-time hyperglycemia and to compare the difference in glucagon secretion when mealtime bolus insulin is given before the meal versus after the meal with the objective of understanding factors that contribute to the peak post-prandial blood glucose and AUC of blood glucose after a mixed meal in this target population.

Hypothesis

1. Patients with higher glucagon responses to a mixed meal stimulus will have higher peak post-prandial glucoses and greater AUC of post-prandial glucose.
2. Bolus dose insulin given pre-meal (20 min before meal) will result in lower peak post-prandial glucose, lower AUC and lower post-prandial glucagon levels
3. Bolus dose insulin given post-meal (20 min after meal) will result in higher peak post-prandial glucoses, higher AUC of post-meal glucose and higher glucagon levels
4. There will be a correlation between peak post-prandial glucagon response and post-meal glucose AUC, 0 to 180 minutes.

Research Plans The study will be conducted in the (Intensive Research Unit, part of the CTSA) Diabetes Center at Barnes Jewish Hospital/Washington University in St Louis.

Study Visits

* Screening will be done over the phone and with review of medical records if the required labs have been done in the past 6 months
* Visits A and B will be performed in random order
* Demographics, review of diabetes history, medications and allergies will be recorded at the first study visit. Insulin doses and effectiveness of current carbohydrate ratio will be evaluated and recorded. Mealtime insulin doses will be established at the first study visit.
* Mealtime insulin will be given via injection by a study nurse to standardize the administration procedure.
* Vital signs, height and weight will be done at each visit
* C-peptide will be checked with the fasting labs at the first study visit
* Baseline glucose should be 80 to 140 mg/dl. In case baseline glucose is not in the target range, the study visit will be rescheduled.
* Whole blood will be collected in vacutainers via an indwelling peripheral venous catheter with nursing supervision.
* Samples will be deidentified before sending to the laboratory.
* No genetic testing will be performed.

Visit A

* Glucose levels done fasting, 30, 60, 120, and 180 minutes
* Glucagon levels done fasting, 30, 60, 120, and 180 minutes
* Usual insulin dose will be administered 20 minutes prior to a mixed meal challenge with Ensure Plus*

Visit B

* Glucose done fasting, 30, 60, 120, and 180 minutes
* Glucagon levels done fasting, 30, 60, 120, and 180 minutes
* Usual insulin dose will be administered 20 minutes after the mixed meal challenge with

Ensure Plus*

*Ensure Plus (Abbott Nutrition) at 6cc/kg (max 360 cc), content per 100 ml: carbohydrate 21.5 grams, protein 5.5 grams, with nursing supervision.

Laboratory Measures:

Core Laboratory for Clinical Studies at Washington University (https://research.wustl.edu/core-facilities/core-laboratory-clinical-studies, CLCS) will measure glucose on the Roche cobas c510 platform using Roche's coupled enzymatic assay (hexokinase, glucose-6-phosphoate dehydrogenase). The rate of NADPH formation is directly proportional to glucose concentration and measured photometrically. The interday imprecision is typically <2.0% CV. CLCS will also measure C-peptide on the Roche cobas e601platform using Roche's sandwich electrochemiluminescence immunoassay. In this assay a biotinylated monoclonal C-peptide-specific antibody and a monoclonal C-peptide-specific antibody labeled with a ruthenium complex bind to C-peptide to form the sandwich. Then, using streptavidin-coated microparticles, the complex is drawn into the measuring cell and remains while unbound material is washed away. Application of a voltage to the electrode induces chemiluminescent emission that is measured by the instrument. Between run precision typically ranges from 1.9 - 2.7% CV.

Glucagon is measured using a radioimmunoassay kit from Millipore. This is a competitive immunoassay which uses I-125 labeled glucagon and a glucagon-specific antibody. Its stated inter-assay precision is 12% CV. Typical within-run precision is 2.0 - 3.0 % CV in our hands.

Methods of Data Analysis Data analysis will be performed using STATA 15.1 for Windows (StataCorp LP, College Station, Texas, United States). The sample size calculation assumes that the peak postprandial glucose will increase by 80 +/-20 mg/dl in the pre-meal insulin group and 140 +/-20 mg/dl in the post-meal group. So, the expected mean peak of postprandial glucose will be up to 220 mg/dL for Visit A and mean peak postprandial glucose will be up to 280 mg/dL for Visit B. The sample size will have 80% power to detect a difference between groups at p<0.05. We have assumed correlation between visits A and B of 0.5. The sample size was corrected by an anticipated loss of follow up of 10% of the participants. The calculated sample size is 10 participants with full data sets available for 8 participants. The study randomization is designed as follows: 5 participants will first attend Visit A, and then Visit B. The 5 remaining participants will first attend Visit B and then Visit A. AUC of post-prandial glucose and glucagon and maximum postprandial peak of glucose and glucagon will be analyzed by using paired T student. Relationships between variables were assessed by a Spearman's correlation test.

ELIGIBILITY:
Inclusion Criteria:

* 10 persons with T1D for >5 years age >18.
* HbA1c <9.5%
* Patients using either MDI or insulin pumps will be included.
* Patients using CGM will continue the use during the study, however glucoses will be measured by laboratory methods.
* Persons of all races, ethnicity and genders will be included
* Participants should have normal hemoglobin, hematocrit and eGFR >60 ml/min/1.73m2.

Exclusion Criteria:

* Persons with type 2 diabetes, monogenic diabetes, pancreatic diseases.
* Pregnancy, prisoners, other vulnerable populations or persons unable to understand the protocol and provide written informed consent.
* Persons who take daily steroids, any route, for any purpose

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet McGill, MD, Principal Investigator — Wash. Univ. School of Medicine
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cryer PE. Minireview: Glucagon in the pathogenesis of hypoglycemia and hyperglycemia in diabetes. Endocrinology. 2012 Mar;153(3):1039-48. doi: 10.1210/en.2011-1499. Epub 2011 Dec 13. PMID 22166985
- [Background] Cooperberg BA, Cryer PE. Insulin reciprocally regulates glucagon secretion in humans. Diabetes. 2010 Nov;59(11):2936-40. doi: 10.2337/db10-0728. Epub 2010 Aug 23. PMID 20811038
- [Background] Vergari E, Knudsen JG, Ramracheya R, Salehi A, Zhang Q, Adam J, Asterholm IW, Benrick A, Briant LJB, Chibalina MV, Gribble FM, Hamilton A, Hastoy B, Reimann F, Rorsman NJG, Spiliotis II, Tarasov A, Wu Y, Ashcroft FM, Rorsman P. Insulin inhibits glucagon release by SGLT2-induced stimulation of somatostatin secretion. Nat Commun. 2019 Jan 11;10(1):139. doi: 10.1038/s41467-018-08193-8. PMID 30635569
- [Background] Schiffrin A, Suissa S, Weitzner G, Poussier P, Lalla D. Factors predicting course of beta-cell function in IDDM. Diabetes Care. 1992 Aug;15(8):997-1001. doi: 10.2337/diacare.15.8.997. PMID 1505333
- [Background] Yosten GLC. Alpha cell dysfunction in type 1 diabetes. Peptides. 2018 Feb;100:54-60. doi: 10.1016/j.peptides.2017.12.001. PMID 29412832
- [Background] Porksen S, Nielsen LB, Kaas A, Kocova M, Chiarelli F, Orskov C, Holst JJ, Ploug KB, Hougaard P, Hansen L, Mortensen HB; Hvidore Study Group on Childhood Diabetes. Meal-stimulated glucagon release is associated with postprandial blood glucose level and does not interfere with glycemic control in children and adolescents with new-onset type 1 diabetes. J Clin Endocrinol Metab. 2007 Aug;92(8):2910-6. doi: 10.1210/jc.2007-0244. Epub 2007 May 22. PMID 17519307
- [Background] Brown RJ, Sinaii N, Rother KI. Too much glucagon, too little insulin: time course of pancreatic islet dysfunction in new-onset type 1 diabetes. Diabetes Care. 2008 Jul;31(7):1403-4. doi: 10.2337/dc08-0575. PMID 18594062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one participant enrolled. Each participant acted as their own control. One participant completed arm A:B.
Groups:
- A (Pre-prandial Insulin Administration) : B (Post-prandial Insulin Administration): Visit 1: will receive short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal. Visit 2: will receive short action insulin (Humalog, Lispro, etc.) with the same regiment patient was using at home 20 minutes after the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
- B: (Post-prandial Insulin Administration): A (Pre-prandial Insulin Administration): Visit 1: will receive short action insulin (Humalog, Lispro, etc.) with the same regiment patient was using at home 20 minutes after the meal Visit 2: will receive short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
Period: Overall Study
Arm/Group | A (Pre-prandial Insulin Administration) : B (Post-prandial Insulin Administration) | B: (Post-prandial Insulin Administration): A (Pre-prandial Insulin Administration)
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Trial was terminated due to COVID pandemic and loss of funding.
Groups:
- A (Pre-prandial Insulin Administration) / (Post-prandial Insulin Administration): Visit 1: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal. Visit 2: will give short action insulin (Humalog, Lispro, etc.) with the same regiment patient was using at home 20 minutes after the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
- B (Post-prandial Insulin Administration) / (Pre-prandial Insulin Administration): Visit 1: will give short action insulin (Humalog, Lispro, etc.) with the same regiment patient was using at home 20 minutes after the meal; Visit 2: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
- Total: Total of all reporting groups
Arm/Group | A (Pre-prandial Insulin Administration) / (Post-prandial Insulin Administration) | B (Post-prandial Insulin Administration) / (Pre-prandial Insulin Administration) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
HbA1c [Number; unit: percent of glycated hemoglobin] | 8.2 |  | 8.2
cPeptide [Number; unit: ng/mL] | 0.003 |  | 0.003
A: Baseline fasting blood glucose (BG) [Number; unit: mg/dL] | 193 |  | 193
Visit B - Baseline Fast Blood Glucose [Number; unit: mg/dL] | 171 |  | 171

OUTCOME MEASURES:

1. Primary Outcome: AUC Postprandial Glucagon
Description: Glucagon levels done fasting, 30, 60, 120, and 180 minutes
Time Frame: 4 hours
Population: Study was delayed and then terminated due to COVID pandemic, funding was lost so primary analysis was not performed.
Groups:
- Pre-prandial Insulin Administration: Pre-prandial insulin: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
- Post-prandial Insulin Administration: Post-prandial insulin: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min post the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
Arm/Group | Pre-prandial Insulin Administration | Post-prandial Insulin Administration
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: AUC Postprandial Glucose
Description: * Glucose done fasting, 30, 60, 120, and 180 minutes
  * Glucagon levels done fasting, 30, 60, 120, and 180 minutes
  * Usual insulin dose will be administered 20 minutes before or after the mixed meal challenge with Ensure Plus*
Time Frame: 4 hours
Measure: Number; unit: mg/dL
Groups:
- Post-prandial Insulin Administration:: Post-prandial insulin: will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min post the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
Arm/Group | Pre-prandial Insulin Administration | Post-prandial Insulin Administration:
Number analyzed (Participants) | 1 | 1
mg/dL
  30 minutes | 245 | 278
  60 minutes | 279 | 316
  120 minutes | 310 | 274
  180 minutes | 301 | 249

ADVERSE EVENTS:
Time Frame: 60 days
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Pre-prandial Insulin: Will give short acting insulin (Humalog, Lispro, etc) with the same regimen patient was using at home 20 min prior the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
- Post-prandial Insulin: Will give short action insulin (Humalog, Lispro, etc.) with the same regiment patient was using at home 20 minutes after the meal.
  Insulin: to give pre-prandial and post-prandial insulin (will use patient insulin dose patient use at home) to patients with T1D and evaluate the response of post-prandial glucagon and post-prandial hyperglycemia.
Arm/Group | Pre-prandial Insulin | Post-prandial Insulin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Study was terminated before completion due to COVID pandemic and loss of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT04079881/Prot_SAP_000.pdf